CLINICAL TRIAL: NCT01677351
Title: Assessment of the Effect of Clonidine on Pain, Arterial and Intraocular Pressure and Arrhythmias for Cataract Surgery
Brief Title: Assessment of the Effect of Clonidine for Cataract Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Ellen de Queiroz Santiago, medical resident, principal investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP 0609/01-clonidine
Record Dates: First submitted 2012-08-01; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Pain; Arrythmia
Keywords: clonidine; cataract surgery; arrythmia; anesthesic medication
MeSH Terms: conditions — Pain; Arrhythmias, Cardiac | interventions — Clonidine; Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 2: clonidine 4mcg.kg (Active Comparator): this group (group 2) will receive 4mcg.kg-1 of clonidine 20 minutes before surgery.
  Interventions: Drug: Clonidine
- Group 1: sterile saline solution (Placebo Comparator): this group (Group 1) will receive a sample injection of sterile saline solution 20 minutes before surgery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Clonidine — 4 mcg.kg-1, 20 minutes before cataract surgery
  Other Names: cataract surgery; anesthesic drugs
  Arms: group 2: clonidine 4mcg.kg
Drug: placebo
  Arms: Group 1: sterile saline solution

SUMMARY:
Clonidine, an agonist for alfa2 pre-synaptic, has been shown to be an effective adjuvant therapy for acute postoperative pain and has been shown an effect in sedative, intra-ocular and blood pressure and arrhythmias.The objective of this study is evaluating the analgesic effect of clonidine and its repercussion on arterial and intraocular pressure and arrhythmias for cataract surgery.

DETAILED DESCRIPTION:
After approved by the Ethical Committee and signed informed consent, 40 patients aged from 40 until 80 years undergoing cataract extraction will be randomized in two groups. Exclusion criteria will be myocardial ischemia, psychiatric disease, chronic pain, drugs dependency, chronic use of beta-blockage channel drugs. Group 2, patients will receive a single dose of 4mcg.kg-1 of clonidin2, 20 minutes before the surgical incision; group 1, patients will receive a sterile saline solution dose. Pain intensity will be assessed with the numeric rating scale. The antiarrythmic effect will be assessed with the continuous measure by Holter. The number of patients was calculated by Instat Graph® program. To detect difference in pain intensity of 3 between the groups by NRS, with 95% of power (estimated SD= 2.0), when the alpha level is set at 0.05, the sample should be of 20. Statistical analyses will be performed with parametric and nonparametric tests, considering the variety studied. The statistical program that will be utilized is Instat Graph®.

ELIGIBILITY:
Inclusion Criteria:

* cataract surgery
* topical anesthesia

Exclusion Criteria:

* myocardial ischemia
* psychiatric disease
* chronic pain
* drugs dependency
* use of beta-blockage channel drugs

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
intensity of pain | 30 minutes before surgery, during the surgery
  Pain intensity will be assessed by numeric rating scale.

SECONDARY OUTCOMES:
intraocular pressure | 30 minutes and during the surgery
  Intra-ocular pressure will be assessed with a manual tonometer of perkins.

OTHER OUTCOMES:
antiarrythmic effect | 30 minutes before surgery and during the surgery
  The antiarrythmic effect will be assessed with the continuous measure by Holter.
blood pressure | 30 minutes before and during the surgery
  Blood pressure will be monitorized with a multiparameter monitor, a non-invasive measure.

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, Study Chair, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Santiago AE, Issy AM, Sakata RK. Effects of preoperative intravenous clonidine in patients undergoing cataract surgery: a double-blind, randomized trial. J Ophthalmol. 2014;2014:346549. doi: 10.1155/2014/346549. Epub 2014 Sep 2. PMID 25276415